CLINICAL TRIAL: NCT05076214
Title: A Randomised Multicentre Study Comparing Vigorous Group Aerobic Exercise vs. Group Leisure Activities for Mild to Moderate Depression in Adolescents
Brief Title: Aerobic Versus Leisure Group for Adolescents With Depression
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Lund University Hospital (Other)
Collaborators: Region Halland (Other); Halmstad University (Other); Karolinska University Hospital (Other); The Rydberg Laboratory for Applied Sciences, Halmstad, Sweden (Unknown); Region Skane (Other); PRIMA Barn- och Vuxenpsykiatri AB (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: LundUH_multicentre
Record Dates: First submitted 2021-09-21; First posted 2021-10-13 (Actual); Last update posted 2025-03-26 (Actual); Status verified 2025-03

CONDITIONS: Depressive Disorder, Major
Keywords: adolescent; depression; exercise intervention; leisure intervention; biomarker; cost evaluation; qualitative
MeSH Terms: conditions — Depressive Disorder, Major; Depression | interventions — Exercise; Population Groups

STUDY DESIGN:
Intervention Model Description: Randomised controlled study
Who Masked: Outcomes Assessor
Masking Description: The patient is at the follow-up interview instructed not to disclose any information about mode of treatment. All interviews are recorded.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Aerobic exercise in group (Experimental): The patients will participate in aerobic group exercise for 60 minutes three times a week for 12 weeks with continuous heart rate monitoring. The sessions will be held in a small gym under supervision of a personal trainer.
  The group training session will begin with a 3-5 minutes check-in round followed by a warm-up to increase heart rate including balance tasks and dynamic stretching for 10-15 minutes. Every third session will be pure aerobic training, every third session will be strengthening exercises designed to also increase heart rate, and every third session will be a mixed session of both aerobic and strength exercises. All major muscle groups will be used at each session. Interval training with gradually increased intensity throughout the program will be applied
  Interventions: Behavioral: Aerobic exercise in group
- Leisure activities in group (Active Comparator): The control group will receive leisure activity in a group setting for one hour three times a week for 12 weeks. The sessions will be held at the same weekdays and about the same hours as the exercise group sessions. The same group leaders as in the exercise sessions will participate in leisure sessions and will support the adolescents through reminders and reassurance before and during the sessions to enhance adherence. The sessions will start with a check in on feelings, recent events and difficulties (i.e. supportive listening but not any interventions) followed by non heart rate increasing activities, such as playing games or cards together.
  Interventions: Behavioral: Leisure activities in group

INTERVENTIONS:
Behavioral: Aerobic exercise in group — The goal with every new week should be making every workout a little bit harder than the week before.
  Strength sessions
  Week 1- 6: 12-18 repetitions (reps) x 2 set per exercise and muscle 30 seconds (s) rest between exercise Week 7-12: 10-12 reps x 3 set per exercise and muscle 20 s rest between exercises Adding weight with gym equipment or changing body position in the exercises to succeed with the rep scheme and making it harder as the group develop their physical and mental ability.
  Conditioning sessions
  Week 1- 6: 75 seconds work time x 1 set per exercise 30 seconds of rest between exercises Week 7-12: 50 seconds work time x 2 set per exercise 20 seconds of rest between exercises Mixed sessions
  Week 1- 6: 35 s work time per exercise 25 s rest between exercises x 2 rounds Week 7-12: 45 s work time per exercise 15 s rest between exercises x 2 rounds
  Arms: Aerobic exercise in group
Behavioral: Leisure activities in group — The control group will receive leisure activity in a group setting for one hour three times a week for 12 weeks. The sessions will be held at the same weekdays and about the same hours as the exercise group sessions. The same group leaders as in the exercise sessions will participate in leisure sessions and will support the adolescents through reminders and reassurance before and during the sessions to enhance adherence. The sessions will start with a check in on feelings, recent events and difficulties (i.e. supportive listening but not any interventions) followed by non heart rate increasing activities, such as playing games or cards together
  Arms: Leisure activities in group

SUMMARY:
The aim is to evaluate aerobic group exercise versus leisure group activities in adolescents with mild to moderate depression.

Primary outcome is Children's Depression Rating Scale - Revised (CDRS-R). Secondary outcomes are Clinical Global Impressions - Severity and Improvement scales (CGI), self-reported Quick Inventory of Depression Symptomatology (QIDS- A17-SR), the self-reported Outcome Rating Scale (ORS), clinician rated Children Global Assessment Scale (C-GAS), aerobic capacity (VO2max), muscular strength, body, Body Mass Index (BMI), presence or activity of selected biological markers of neuroprotection and neuroinflammation in blood samples and a cost evaluation rated by parents with Trimbos/iMTA questionnaire for Costs associated with Psychiatric Illness - Child version (Tic-P) and the Child Health Utility (CHU9D) to facilitate estimation of Quality Adjusted Life Years. Further objectives are qualitative interviews to explore adolescents' experiences of the intervention as well as how their health and lifestyle are influenced and a validation of QIDS- A17-C and QIDS- A17-SR versus CDRS-R will be performed.

DETAILED DESCRIPTION:
Depression is common in adolescence and prevalence is increasing. It is a major cause of disability worldwide and contributes to lower educational achievements, increased risk of substance abuse, suicide and cardiovascular disease. The effect of evidence based treatments with antidepressants or psychotherapy such as cognitive behavioural therapy (CBT) or interpersonal therapy (IPT) are modest. Selective serotonin uptake inhibitors (SSRIs) have shown effect on depression in children and adolescents, but the effect is often insufficient.

Aerobic exercise seems to have effect on depression in adolescents but studies have several shortcomings. Recruitment was mostly in non-clinical or primary care facilities, results are heterogeneous and adequate control groups are lacking. More data on qualitative, cost-effectiveness and biomarker aspects are clearly warranted.

OBJECTIVES:

Primary objective: To evaluate aerobic group exercise versus leisure group activities on clinician rated depression symptoms among adolescents in child and adolescent outpatient care with mild to moderate depressive disorder by measuring changes in Children's Depression Rating Scale- Revised (CDRS-R) after the intervention at 13 weeks from baseline.

Secondary objectives: To evaluate change in CDRS-R also at 26 weeks after baseline, i.e. after a period of no active intervention. Other secondary objectives are at both 13 and 26 weeks clinician rated Clinicial Global Impression - Severity (CGI-S) and Clinical Global Impression - Improvement scale (CGI-I) and function with Children Global Assessment Scale (C-GAS), self-rated symptoms (QIDS-A17-SR) and function with the Outcome Rating Scale (ORS), aerobic capacity measured by a submaximal aerobic capacity test, muscular strength measured by the isometric mid-thigh pull strength test, a hand grip strength test and muscular endurance by the one-leg sit-to-stand test, and body composition with a bioelectrical impedance analysis and presence or activity of selected biological markers of neuroprotection and neuroinflammation in blood samples.

Moreover, the investigators will assess cost-effectiveness. Also to explore adolescents' experiences of the intervention as well as how their health and lifestyle are influenced by the intervention through qualitative interviews. Finally, to validate QIDS- A17-C and QIDS-A17-SR against CDRS-R.

DESIGN: The study will be a multi centre randomised pilot study that will include 122 adolescents with ongoing mild to moderate depression after three or more vlinical visits. Participants will be randomised to receive 12 weeks of either aerobic group exercise or leisure group activities at a ratio of 1:1. Adolescents allocated to leisure activities will get the opportunity to participate in aerobic exercise after the evaluation at 26 weeks.

Control group justification: Leisure activities in a group setting to control for the possible effect on social interaction and behavioural activation.

Study setting: The study will be conducted at the child and adolescent psychiatric clinic in Halmstad, Kungsbacka, Stockholm and Malmö, Sweden. The sites are the only providers of specialised care for adolescent depression in their geographical areas. Outcome variables are assessed by communicating with patients on smart phones. Research interviews will be recorded video calls, and self-rated measures collected electronically.

POWER ANALYSIS: The statistical power is based on a pilot study (id: 2020-03364) with a beta of 80% and an alpha of 0.05 and a 25% attrition arriving at 122 participants.

DATA COLLECTION: QIDS-A17-SR and K-SADS-PL with the adolescent and parent will be conducted at the clinics before baseline. CDRS-R, QIDS-A17-C and CGAS at baseline, 13 weeks, 26 weeks and one- year follow up assessment will be conducted through a recorded video call. At baseline, 13 weeks, 26 weeks and at one-year parents will web-based fill in Tic-P for costs and participants fill in the CHU9D for quality of lifePatients fill out a web based questionnaire with QIDS-A17-SR and ORS every two weeks during the 12 weeks intervention period and monthly during the follow-up until one year.

SCREENING AND RECRUITMENT PROCEDURES: The investigators will from outpatient clinics recruit patients diagnosed with depression and who have had at least three visits and thus most likely have received some basic psychosocial interventions. The patients will be identified through a scanning of the outpatient computer system.

RANDOMISATION, ENROLMENT AND MASKING: Participants will be randomised at a ratio of 1:1 to aerobic group exercise or group leisure activities. Sealed envelopes with randomisation numbers will be stored in a locked cabinet. Randomisation will occur for each site to arrive at equally sized groups if full inclusion is not possible within the set time frame.

The investigators Tina Cronqvist (TC) and Rebecca Mortazavi (RM) conducting the baseline, 13 and 26 week evaluation will be blind to treatment allocation. The outcome measures are identical for the two groups, ensuring that the assessors remain blind. Participants will be reminded at the start of each interview not to reveal their arm of allocation. To measure blinding integrity, the assessor will record whether the participating patients inadvertently reveal their group allocation. If the patient disclose treatment arm, this part of the recording will be deleted in a copied version and the interview is rated by the other rater. At the one-year open follow up, all patients have had the opportunity to exercise and the evaluation is unblinded.

RATER TRAINING: TC and RM will get instructions and perform CDRS-R supported by an experienced user of CDRS-R including rating and discussions of four recorded videos.

BASELINE ASSESSMENTS: Clinician video evaluation: CDRS-R, QIDS-A17-C, CGI-I and C-GAS will be conducted through a recorded video call. Inter rater test will be performed between RW, TC and PI on ten CDRS-R, C-GAS and QIDS-A17-C from baseline.

Self-reported web based: QIDS-A17-SR, CHU9D and ORS.

Parent cost evaluation web based with the Treatment Inventory of Costs in Psychiatric Patients (Tic-P).

Measures at site: aerobic capacity, muscular strength and body composition.

Blood sampling to be stored in a freezer.

RECURRENT EVALUATIONS: QIDS-A17-SR and ORS will be filled in every two weeks during the 12 week active intervention and monthly during the remainder of the study year. After two weeks of intervention patients will also fill in questions on safety, side effects and treatment credibility.

13 WEEK EVALUATION Clinician video evaluation: CDRS-R, CGI and C-GAS Self-reported web based: QIDS-A17-SR, CHU9D and ORS Parent rated and web-based cost evaluation with Tic-P Qualitative interviews with participants according to interview guide Anthropometric measures at site: height, weight, aerobic capacity, muscular strength and body composition.

Blood sampling

26 WEEK EVALUATION Clinician video evaluation: CDRS-R, CGI and C-GAS Self-reported web based: QIDS-A17-SR, CHU9D and ORS Parent rated and web-based cost evaluation with Tic-P

ONE YEAR EVALUATION: Identical to baseline assessments but also qualitative interviews with patients and parents.

END OF TRIAL: The trial will end when the final data from the one-year follow up has been collected for the last patient.

PARTICIPANT WITHDRAWAL: Participants are free to withdraw from the trial at any point. After the withdrawal, participants will not be requested to complete any measures, but will be asked to provide non-obligatory feedback regarding their reason for withdrawal Once participants have withdrawn from the trial, it will not be possible to re-enter or resume treatment. Withdrawn patients will not be replaced in the trial. Patients will be asked to have their data withdrawn.

CONCOMITANT INTERVENTIONS: Medication for depression is required to have been stable for four weeks prior to inclusion. Medications with stimulants or neuroleptics need to have been stable for two weeks. Additionally, the participants are encouraged not to alter medication or receive any psychological treatment until after the 26 week evaluation. Visits for safety evaluations, school-planning and to issue parental child-sick leave are permitted.

DATA MANAGEMENT: All aspects of data management of the trial will comply with the General Data Protection Regulation (GDPR). Notes will be made in the clinical records.

STATISTICAL ANALYSES: Demographic data will be summarised using descriptive statistics. T-tests will be performed to investigate if missing data at the three follow up measures can be considered as missing at random (MAR). More specifically, baseline scores for the participants with missing data will be compared with baseline scores for participants with complete data on all outcome variables. Multiple imputation using the predictive mean matching approach will be used to replace missing values for CDRS-R, using data from the QIDS-A-17 self rating scales, baseline scores on the CDRS-R and relevant patient characteristics (e.g., age, sex) as input variables in the model. For more information about this approach see van Ginkle et al. (2020). Data analysis will be conducted using linear mixed models (LME) to analyse change in outcome variables following the interventions. Time will be specified as a fixed effect parameter. Random effects parameters are in intercept and linear slope terms. An unstructured covariance matrix will be used to account for within patient correlation across time. A two-sided 95% confidence interval will be used to assess the treatment effect, with statistical significance determined if the confidence interval does not include zero. Cohen's f will be used as the effect size measure for the statistical tests. The main analysis will be performed by an extern statistican, blind to randomisation.

ADVERSE EVENTS:

Serious Adverse Event (SAE) is any unfortunate occurrence that:

results in death is life-threatening requires hospitalisation results in persistent or significant disability or incapacity is otherwise considered medically significant by the investigator

Suspected Unexpected Serious Adverse Reaction (SUSAR) is any SAE that is deemed to be:

related to the trial intervention AND unexpected AND not listed in the protocol as an expected adverse event of the intervention.

The investigators have considered the following events as possible adverse events:

Increased depressive symptoms. Suicide attempt. Increased stress due to time consuming sessions and transportation. Injuries due to exercise. The investigators also have to consider that adverse events may also be symptoms of the underlying depressive disorder, rather than the intervention itself.

The assessment of the relationship between adverse events and the administration of the treatment is a decision based on all available information. The final decision is taken by the PI. If the event is a result of the administration of any of the research procedures then it will be classified as related.

If the event has been listed in the protocol as an expected side effect of the intervention then the event will be classified as expected. If the event is not listed then it will be classified as unexpected.

All adverse events will be noted by the trial coordinator in a specific log (including date, recorded clinical symptoms, and a brief description of the event). SAEs and SUSARs will be recorded in the trial coordinator's log. Appropriate action will be taken in the case of SAE and SUSAR, making sure the participant will get in contact with suitable health care services. Events will be considered as potentially treatment-related up to the 13 weeks evaluation, where the reporting of adverse events will terminate.

Notification of serious breaches to Good Clinical Practice (GCP) and/or the protocol

DATA SHARING: The investigators will not share trial data with other researchers around the world.

ETHICAL CONSIDERATIONS: The study is approved by the Swedish Ethical Review Authority (2021-05307-01). All patients and parents will be provided by oral and written information about the study. Informed consent in writing will be provided from patients and parents to participants below 15 years of age.

Participants randomised to leisure activities will get the opportunity to exercise after 26 weeks, ensuring all participants are offered the active treatment.

IMPLICATIONS: Aerobic group exercise can, if shown to be effective, become a recommended treatment option for major depressive disorder in adolescents either alone or as an addition to present treatment options such as cognitive behavioural therapy and antidepressants.

ELIGIBILITY:
Inclusion Criteria:

* DSM-5 mild to moderate depression
* who have received evaluation and basic psychosocial interventions for 4-8 weeks (minimum three visits) without response, i.e. not achieved improvement by at least 50 % as assessed from clinical records

Exclusion Criteria:

* Severe depression
* Eating disorder
* High risk for suicide
* Intellectual disability
* Actual physical activity the last four weeks meeting the level for sustained health by American College of Sports Medicine, i.e. at least 150 min per week of moderate intensity or 75 min per week of high intensity38
* Adjustment of antidepressant medication within the last four weeks or stimulants the last two weeks
* Chronic somatic illness precluding exercise
* In need of interpreter
* Social circumstances interfering with a regular exercise schedule
* Concomitant psychotherapy

Ages: 13 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 122 (Estimated)
Dates: Start 2022-02-28 (Actual); Primary Completion 2025-06-10 (Estimated); Study Completion 2026-03-10 (Estimated)

PRIMARY OUTCOMES:
Change in Children's Depression Rating Scale- Revised (CDRS-R) | After intervention (at 13 weeks = primary endpoint) but also at 26 weeks (still blinded)and at follow-up (at 52 weeks, non-blinded)
  Clinician administered interview about symptoms of depression, range 17 (best) - 113 (worst)

SECONDARY OUTCOMES:
Change in Quick Inventory of Depressive Symptomatology - Adolescent version, Self Report (QIDS-A17-SR) | Every two weeks during the 12 week intervention and monthly during the following year.
  Self report form about symptoms of depression, range 0 (best) - 27 (worst)
Clinical Global Impression - Severity | After intervention (at 13 weeks), at 26 weeks and at follow-up (at 52 weeks)
  Clinician determined overall measure of severity pf psychopathology, values ranging from 1 (normal and best) to 7 (among the most extremely ill patients and worst)
Clinical Global Impression - Improvement | After intervention (at 13 weeks), at 26 weeks and at follow-up (at 52 weeks)
  Clinician determined overall measure of change from initiation of treatment, values ranging from 1 (very much improved and best) to 7 (very much worse and worst)
Change in Children Global Assessment Scale (C-GAS) | After intervention (at 13 weeks), at 26 weeks and at follow-up (at 52 weeks)]
  Clinician administered interview about psychosocial function, 1(worst) - 100 (best
Change in Outcome Rating Scale (ORS) | Every two weeks during the 12 week intervention and monthly during the following year.
  Self report form about psychosocial function, range 1 (worst) - 100 (best)
Change in Aerobic capacity | After intervention (at 13 weeks) and at follow-up (at 52 weeks)
  Submaximal and maximal aerobic capacity test, measured as Oxygen consumption (ml) / weight (kg) x time (minute), range typically about 20 (lowest) - about 60 (highest)
Change in Muscular strength | After intervention (at 13 weeks) and at follow-up (at 52 weeks)
  Change in Isometric mid-thigh pull strength test (kg), a hand grip strength test (kg)
Change in muscular endurance | After intervention (at 13 weeks) and at follow-up (at 52 weeks)
  time to repeat 5 one-leg sit-to-stand test (seconds, lower value indicates increased muscular endurance))
Change in body composition | After intervention (at 13 weeks) and at follow-up (at 52 weeks)
  body composition with a bioelectrical impedance analysis (resistance in Ohm, lower value indicates increase in muscle and higher value increase in fat)
Change in Brain Derived Neurotrophic Factor (BDNF) in blood samples | After intervention (at 13 weeks) and at follow-up (at 52 weeks)
  Biomarker BDNF for neuroprotection (higher value is better) and associated binding proteins.
Change in Kynerunic Acid (KYNA)/3HK75 in blood samples | After intervention (at 13 weeks) and at follow-up (at 52 weeks)
  Biomarker KYNA/3HK75 for neuroprotection (higher value is better) and associated binding proteins.
Change in Kynerunic Acid (KYNA) / Quinolinic Acid (QUIN)75 in blood samples | After intervention (at 13 weeks) and at follow-up (at 52 weeks)
  Biomarker KYNA/QUIN75 for neuroprotection (higher value is better) and associated binding proteins.
Change in Kynerunic Acid (KYN-ACID)75 in blood samples | After intervention (at 13 weeks) and at follow-up (at 52 weeks)
  Biomarker KYN-ACID75 for neuroprotection (higher value is better) and associated binding proteins.
Change in C-reactive Proteins (CRP) in blood samples | After intervention (at 13 weeks) and at follow-up (at 52 weeks)
  Biomarker CRP for neuroinflammation (lower value is better) and associated binding proteins.
Change in Interleukin (IL)-6 in blood samples | After intervention (at 13 weeks) and at follow-up (at 52 weeks)
  Biomarker IL-6 for neuroinflammation (lower value is better) and associated binding proteins.
Change in Soluble Interleukin (SIL)-2 receptor in blood samples | After intervention (at 13 weeks) and at follow-up (at 52 weeks)
  Biomarker SIL-2 receptor for neuroinflammation (lower value is better) and associated binding proteins.
Change in Tumor Necrosis Factor (TNF)-alpha in blood samples | After intervention (at 13 weeks) and at follow-up (at 52 weeks)
  Biomarker TNF-alpha for neuroinflammation (lower value is better) and associated binding proteins.
Change in Insulin-like Growth Factor (IGF)-1 in blood samples | After intervention (at 13 weeks) and at follow-up (at 52 weeks)
  Biomarker IGF-1 for neuroinflammation (lower value is better) and associated binding proteins.
Change in costs with the Treatment Inventory of Costs in Psychiatric Patients (Tic-P) | After intervention (at 13 weeks), at 26 weeks and at follow-up (at 52 weeks)
  Change in costs for consumption of health care, costs associated with mental illness and production loss among parents due to psychiatric problems in the child concerning the previous four weeks compared to the four weeks before start of intervention (in Swedish crowns), lower cost is better.
Change in quality of life through Child Health Utility 9D (CHU9D) | After intervention (at 13 weeks), at 26 weeks and at follow-up (at 52 weeks)
  Change in quality of life on nine dimensions and a composite value ranging from 0 (lowest) to 1 (highest)

CONTACTS AND LOCATIONS:
Locations (4):
- Sweden (4):
  - Region Halland, Halmstad
  - Prima Barn och vuxenpsykiatri AB (Stockholm-Handen), Stockholm
  - PRIMA Barn och vuxenpsykiatri AB (Stockholm-Järva), Stockholm
  - Region Halland, Varberg

IPD SHARING:
Plan to Share IPD: No
The data are shared in a pseodu-anonymised form within the research group but not beyond the research group.

REFERENCES:
- [Background] Mortazavi R, Lalouni M, Grudin R, Serlachius E, Sundberg CJ, Norrbom J, Larsson I, Haglund E, Ivarsson A, Lenhard F, Cronqvist T, Ingemarsson K, Marsell A, Rask O, Jarbin H. Moderate-to-vigorous group aerobic exercise versus group leisure activities for mild-to-moderate depression in adolescents: study protocol for a multicentre randomised controlled trial. BMJ Open. 2022 Jul 12;12(7):e060159. doi: 10.1136/bmjopen-2021-060159. PMID 35820753
- [Background] Jarbin H, Hoglund K, Skarphedinsson G, Bremander A. Aerobic exercise for adolescent outpatients with persistent major depression: Feasibility and acceptability of moderate to vigorous group exercise in a clinically referred sample. Clin Child Psychol Psychiatry. 2021 Oct;26(4):954-967. doi: 10.1177/13591045211000782. Epub 2021 Apr 16. PMID 33858215
- [Result] Mortazavi R, Andersson R, Jarbin H, Larsson I. Empowered and engaged: Group exercise for adolescent depression - perspectives from adolescents, parents and healthcare professionals. SAGE Open Med. 2024 Feb 3;12:20503121231225340. doi: 10.1177/20503121231225340. eCollection 2024. PMID 38313468

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2025-03-16): https://cdn.clinicaltrials.gov/large-docs/14/NCT05076214/Prot_SAP_001.pdf